CLINICAL TRIAL: NCT04452981
Title: A Randomized, Double Blind Sham Controlled Clinical Trial to Evaluate The Efficacy of Vestibular Nerve Stimulation (VeNS), Compared to a Sham Control For Treatment Of Insomnia.
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) as a Treatment for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: University of Ulster (Other); The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UUSS001
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Insomnia; Sleep Disturbance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): The active device utilizes a technology termed vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 1 hour per day.
  Interventions: Device: VeNS
- Sham (Sham Comparator): The sham device looks identical to the active device and interacts with the app in a similar manner to the active device. It will apply some stimulation to a user for a limited period of time (30 seconds), before tapering down to zero over a further 20 seconds, thus creating the impression of an active device. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will be advised to use the device at home for 1 hour per day.
  Interventions: Device: VeNS

INTERVENTIONS:
Device: VeNS — The VeNS device utilizes a technology called galvanic vestibular stimulation (GVS) (sometimes termed vestibular nerve stimulation (VeNS)). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 1 hour per day.

SUMMARY:
Insomnia is known to be one of the most common health concerns in in the general population and has been associated with several health consequences. Medications are known to be effective, and currently serve as the primary treatment for insomnia but their use is limited due to the risk of adverse events. Cognitive Behavioral Therapy (CBT-1) has also been shown to be effective and safer in the treatment of insomnia but presents its own limitations such as the time, cost, and training required. The relationship between vestibular stimulation and sleep continues to be explored, however its usefulness in the treatment of insomnia is still unknown. Vestibular stimulation itself has been shown to be safe across multiple populations. If vestibular stimulation is shown to be effective in the treatment of insomnia, it could serve as a safer alternative to medications. It could also require less cost, time, and training than CBT-1, providing a treatment option that is not only safe and effective, but broadly available to the general population. Consequently this trial seeks to evaluate the efficacy of non-invasive electrical vestibular nerve stimulation as a method of improving sleep quality and quantity, as compared to a sham control, in patients newly diagnosed with insomnia.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent
2. Diagnosed insomnia with ISI of 15 or greater at screening
3. Males or females
4. 18-80 years of age inclusive on starting the study
5. Ability and willingness to complete all study visits and procedures; in particular an agreement to engage with trying to use the device on a daily basis
6. Agreement not to use prescription, or over the counter, sleep medications for the duration of the trial
7. Agreement not to use sleep trackers for the duration of the study (e.g sleep app smart watches)
8. Access to Wi-Fi (to connect iPod to internet)

Exclusion Criteria

1. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears (image from participant required).
2. Previous diagnosis of HIV infection or AIDS (HIV is known to cause a vestibular neuropathy which would prevent VeNS from working)
3. Medication for insomnia (unless regime stable for last 3 months).
4. A history of stroke or severe head injury (as defined by a head injury that required a craniotomy or endotracheal intubation). (In case this damaged the neurological pathways involved in vestibular stimulation).
5. Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.).
6. Pregnancy.
7. Previous use of any VeNS device
8. Participation in other clinical trials sponsored by Neurovalens
9. Have a member of the same household who is currently participating in this study.
10. History of vestibular dysfunction or other inner ear disease as indicated by the following screening questions:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) score | 4 weeks
  To evaluate the effect of the VeNS device, relative to control group on participants with insomnia. ISI is a self-report rating scale assessing the severity of insomnia symptoms (range 0-28) with higher scores indicating a more severe insomnia.

SECONDARY OUTCOMES:
Number of adverse events | 4 weeks
  To evaluate the safety of the VeSTAL device relative to control group, in terms of the occurrence of adverse events.
Quality of life using SF-36 scores | 4 weeks
  To evaluate the effect of the VeNS device, relative to control group, on quality of life. SF-36 is a 36-item short form survey (range 0-100) with higher scores indicating a better quality of life.
Quality of sleep using PSQI | 4 weeks
  To evaluate the effect of the VeNS device, relative to control group, on quality of sleep quantified by change in the PSQI score. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Sittlington, PhD, Principal Investigator — University of Ulster
Locations (2):
- School of Nursing, The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong
- University of Ulster, Coleraine, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be transferred in an encrypted PDF format. Trial staff will be given direction on how to share the trial data and given access to one specific section of a controlled cloud service which is controlled via role based access. Once they have authenticated with the service and the service verifies that they have the correct role to access the system they will be directed to a single webpage within the application where they will be able to upload the encrypted PDF. This PDF is generated on the fly and is therefore not stored in another location that could become compromised. Generating the PDF on the fly means that the source data is extracted from the database, processed and delivered in the context of a single request. These data will be transferred for each subject when they complete participation in the study.

REFERENCES:
- [Derived] Cheung T, Lam JYT, Fong KH, Cheng CP, Xiang YT, Li TMH. Efficacy of electrical vestibular stimulation (VeNS) on adults with insomnia: A double-blind, randomized, sham-controlled trial. Dialogues Clin Neurosci. 2025 Dec;27(1):236-248. doi: 10.1080/19585969.2025.2526547. Epub 2025 Jul 11. PMID 40650353
- [Derived] Cheung T, Lam JYT, Fong KH, Cheng CP, Ho A, Sittlington J, Xiang YT, Li TMH. Evaluating the Efficacy of Electrical Vestibular Stimulation (VeNS) on Insomnia Adults: Study Protocol of a Double-Blinded, Randomized, Sham-Controlled Trial. Int J Environ Res Public Health. 2023 Feb 17;20(4):3577. doi: 10.3390/ijerph20043577. PMID 36834268